CLINICAL TRIAL: NCT00722566
Title: An Open-Label Randomized Study of Subcutaneous and Intravenous VELCADE in Subjects With Previously Treated Multiple Myeloma
Brief Title: A Study of Subcutaneous and Intravenous VELCADE in Patients With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138 MMY 3021
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): VELCADE administered by subcutaneous injection
  Interventions: Drug: VELCADE Administered by subcutaneous injection
- 2 (Active Comparator): VELCADE administered by intravenous infusion
  Interventions: Drug: VELCADE Administered by intravenous infusion

INTERVENTIONS:
Drug: VELCADE Administered by subcutaneous injection — Patients will receive a 1.3mg/meters(squared)/dose of VELCADE on Days 1,4,8, and 11 of a 3-week cycle
  Arms: 1
Drug: VELCADE Administered by intravenous infusion — Patients will receive a 1.3mg/meters(squared) dose of VELCADE on Days 1,4,8, and 11 of a 3-week cycle.
  Arms: 2

SUMMARY:
Randomized, open-label, international, multi-center, Phase 3 study in which patients are randomized to receive VELCADE administered by subcutaneous injection or intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years or older
2. Diagnosis of multiple myeloma
3. Measurable, secretory multiple myeloma defined as serum monoclonal IgG of ≥10 g/L, serum monoclonal IgA or IgE ≥5 g/L, or serum monoclonal IgD ≥0.5g/L; or urine M-protein of ≥200 mg/24 hr
4. Relapse or progression of myeloma following prior systemic antineoplastic therapy.

Exclusion Criteria:

1. Previous treatment with VELCADE
2. More than 3 previous lines of therapy (separate lines of therapy are defined as single or combination therapies that are either separated by disease progression or by a greater than 6 month treatment-free interval)
3. Peripheral neuropathy or neuropathic pain of NCI CTCAE Grade ≥2
4. Any of the following within 3 weeks prior to randomization:

   antineoplastic or experimental therapy, corticosteroid use above 10mg a day (prednisone or equivalent), or plasmapheresis
5. Any of the following within 2 weeks prior to randomization:

   radiation therapy, major surgery (kyphoplasty is not considered major surgery)
6. Prior malignancy other than multiple myeloma diagnosed or treated within the last 2 years, with the exception of completely resected carcinoma in situ or basal/squamous carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Ortho Biotech Oncology Research & Development - Unit of Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (3):
- UZ Brussel Department Medical Oncology Laarbeeklaan 101, Brussels, Belgium
- Hôtel DIEU, Service D'Hématologie Place Alexis RICORDEAU, Nantes, France
- Universitätsklinikum Münster Onkologische Ambulanz West Albert-Schweitzer-Str. 33, Münster, Germany

REFERENCES:
- [Derived] Moreau P, Pylypenko H, Grosicki S, Karamanesht I, Leleu X, Rekhtman G, Masliak Z, Robak P, Esseltine DL, Feng H, Deraedt W, van de Velde H, Arnulf B. Subcutaneous versus intravenous bortezomib in patients with relapsed multiple myeloma: subanalysis of patients with renal impairment in the phase III MMY-3021 study. Haematologica. 2015 May;100(5):e207-10. doi: 10.3324/haematol.2014.118182. Epub 2015 Jan 16. No abstract available. PMID 25596270
- [Derived] Moreau P, Pylypenko H, Grosicki S, Karamanesht I, Leleu X, Grishunina M, Rekhtman G, Masliak Z, Robak T, Shubina A, Arnulf B, Kropff M, Cavet J, Esseltine DL, Feng H, Girgis S, van de Velde H, Deraedt W, Harousseau JL. Subcutaneous versus intravenous administration of bortezomib in patients with relapsed multiple myeloma: a randomised, phase 3, non-inferiority study. Lancet Oncol. 2011 May;12(5):431-40. doi: 10.1016/S1470-2045(11)70081-X. Epub 2011 Apr 18. PMID 21507715

RESULTS

PARTICIPANT FLOW:
Groups:
- VELCADE Subcutaneous: VELCADE 1.3 mg/m^2 administered by subcutaneous injection on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles.
- VELCADE Intravenous: VELCADE 1.3 mg/m^2 administered by intravenous infusion on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles.
Period: Overall Study
Arm/Group | VELCADE Subcutaneous | VELCADE Intravenous
Started | 148 (One patient randomized and not dosed) | 74
Completed | 81 (Completed 8 cycles) | 39 (Completed 8 cycles)
Not Completed | 67 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VELCADE Subcutaneous | VELCADE Intravenous | Total
Number analyzed (Participants) | 148 | 74 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 37 | 111
  >=65 years | 74 | 37 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.96) | 64.0 (12.11) | 64.2 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 27 | 101
  Male | 74 | 47 | 121
Region of Enrollment [Number; unit: participants]
  France | 22 | 14 | 36
  Belgium | 7 | 5 | 12
  Germany | 2 | 4 | 6
  Netherlands | 6 | 4 | 10
  United Kingdom | 6 | 3 | 9
  Ukraine | 51 | 17 | 68
  Russian Federation | 26 | 9 | 35
  Poland | 20 | 7 | 27
  Argentina | 5 | 8 | 13
  India | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Overall Response (Complete Response + Partial Response)
Description: Disease response was measured according to European Group for Blood and Marrow Transplantation (EBMT) criteria with the addition of the response categories of nCR and VGPR.
  Complete response requires disappearance of monoclonal protein from the blood and urine and <5% plasma cells in the bone marrow on at least 2 determinations for a minimum of 6 weeks.
  Partial Response requires ≥50% reduction in serum m-protein for at least 2 determinations at least 6 weeks apart and if present, reduction in 24-hour urinary light chain excretion by either ≥90% or to <200 mg
Time Frame: Over 4 cycles (prior to the addition of dexamethasone)
Population: The response-evaluable population was defined as subjects who received at least 1 dose of study drug and had measurable, secretory multiple myeloma, defined as a serum monoclonal IgG or IgM of ≥10 g/L or a serum monoclonal IgA or IgE ≥5 g/L, or a serum monoclonal IgD of ≥0.5g/L, or urine M-protein of ≥200 mg/24 hours, at study entry.
Measure: Number; unit: Participants
Groups:
- VELCADE Subcutaneuous: VELCADE 1.3 mg/m^2 administered by subcutaneous injection on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles.
- VELCADE Intravenous: VELCADE 1.3 mg/m^2 administered by intravenous injection on Days 1, 4, 8, and 11 of a 3-week cycle for 8 cycles.
Arm/Group | VELCADE Subcutaneuous | VELCADE Intravenous
Number analyzed (Participants) | 145 | 73
Participants | 61 | 31
Statistical Analysis 1: Comparison: VELCADE Subcutaneuous vs VELCADE Intravenous; In this trial, non-inferiority is defined as retaining 60% of the IV (active control) treatment effect as measured by ORR. The non-inferiority hypothesis can be stated as: H0: ORRSC - 0.60 ORRIV <0 vs. H1: ORRSC - 0.60 ORRIV ≥0 (non-inferiority); Test type: Non-Inferiority or Equivalence — Assuming ORRs are 35.5% for both SC and IV, one-sided alpha level of 0.025, and approximately 80% power, approximately 216 subjects (144 SC:72 IV) are needed to show non-inferiority of SC to IV VELCADE; p = 0.00201, Farrrington and Manning; CONOR P. FARRINGTON AND GODFREY MANNING STATISTICS IN MEDICINE, VOL. 9, 1447-1454(1990); ORR_SQ - 0.6 ORR_IV = 16.8, 95% CI 2-sided [6.1 to 27.1]

2. Secondary Outcome: Number of Patients With Complete Response
Description: Disease response was measured according to European Group for Blood and Marrow Transplantation (EBMT) criteria with the addition of the response categories of nCR and VGPR.
  Complete response requires disappearance of monoclonal protein from the blood and urine and <5% plasma cells in the bone marrow on at least 2 determinations for a minimum of 6 weeks.
Time Frame: Over 4 cycles (prior to the addition of dexamethasone)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | VELCADE Subcutaneous | VELCADE Intravenous
Number analyzed (Participants) | 145 | 73
Participants | 9 | 6

ADVERSE EVENTS:
Arm/Group | VELCADE Subcutaneous | VELCADE Intravenous
Serious Adverse Events (participants affected / at risk) | 53/147 | 26/74
Other Adverse Events (participants affected / at risk) | 112/147 | 66/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VELCADE Subcutaneous (N=147) | VELCADE Intravenous (N=74)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Haematemesis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 0
Sudden death (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Hepatitis C (General disorders) | 1 | 0
Herpes Zoster (Infections and infestations) | 2 | 0
Injection site abscess (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 5
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Perianal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0
Paraparesis (Nervous system disorders) | 2 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Peripheral neuropathy motor (Nervous system disorders) | 2 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Neurosis (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Vulval ulceration (Reproductive system and breast disorders) | 1 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VELCADE Subcutaneous (N=147) | VELCADE Intravenous (N=74)
Leukopenia (Blood and lymphatic system disorders) | 29 | 16
Abdominal pain upper (Gastrointestinal disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 21 | 11
Dyspepsia (Gastrointestinal disorders) | 4 | 7
Chills (General disorders) | 6 | 4
Fatigue (General disorders) | 17 | 15
Oedema peripheral (General disorders) | 9 | 6
Nasopharyngitis (Infections and infestations) | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 7 | 7
Weight decreased (Investigations) | 22 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 8
Dizziness (Nervous system disorders) | 10 | 2
Headache (Nervous system disorders) | 5 | 8
Paraesthesia (Nervous system disorders) | 9 | 6
Insomnia (Psychiatric disorders) | 18 | 8
Pruritis (Skin and subcutaneous tissue disorders) | 7 | 2
Rash (Skin and subcutaneous tissue disorders) | 10 | 5
Hypertension (Vascular disorders) | 14 | 3
Chalazion (Eye disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No